CLINICAL TRIAL: NCT03958734
Title: Postprandial Monocyte Maturation and Vascular Dysfunction Following High-Fat Meals: The Impact of Cardiovascular Fitness and Acute Aerobic Exercise - Study 1
Brief Title: Postprandial Monocyte Maturation and Vascular Dysfunction Following High-Fat Meals - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Sigma Xi (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20015510-1
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Risk Factor; Lipemia
Keywords: Vascular Dysfunction
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low physical activity/fitness (Other): Participants will be classified as into low-physical fitness based on self-reported physical activity and cardiorespiratory fitness testing.
  Interventions: Other: High-fat meal
- High physical activity/fitness (Other): Participants will be classified as into high-physical fitness based on self-reported physical activity and cardiorespiratory fitness testing.
  Interventions: Other: High-fat meal

INTERVENTIONS:
Other: High-fat meal — Participants will be given a serving of Marie Callendar's Chocolate Satin Pie to eat over a period of 20 minutes

SUMMARY:
The purpose of this research study is to examine the effect of high-fat meals on the health of blood vessels. In addition, the study will examine how exercise/fitness/physical activity impacts blood vessels after consumption of a high-fat meal.

DETAILED DESCRIPTION:
This is the first in a series of studies examining the impact of high-fat meals on blood vessels. During the preliminary visit of this study, eligible participants' resting metabolic rate, arm flow mediated dilation, and leg flow mediate dilation will be measured. They will complete handgrip and plantar flexion exercise tasks. Finally, they will be given a physical activity monitor to wear for 7 days. At their first visit, participants will eat a high-fat meal and blood will be drawn to measure blood vessel health. They will also repeat the arm flow mediated dilation, leg flow mediate dilation, handgrip, and plantar flexion exercise tests.

ELIGIBILITY:
Inclusion Criteria:

1. college-age: 18-30 years old
2. normal fasting triglyceride (<150 mg/dL) (American College of Sports Medicine Guidelines for Exercise Testing and Prescription, 10th Edition).
3. normal body composition: % body fat, males <25%, females <32% (American College of Sports Medicine Guidelines for Exercise Testing and Prescription, 10th Edition)
4. self-reported engagement in moderate-vigorous intensity physical activity and/or an exercise training regimen OR self-reported low physical activity and no engagement in an exercise training regimen (International Physical Activity Questionnaire)
5. low cardiorespiratory fitness (VO2peak; male: =<45 mL/kg/min; female: =<35 mL/kg/min; categorized as =40th percentile by ACSM Guidelines for Exercise Testing and Prescription, 10th Edition; 44, 45, 46, 47) OR high cardiorespiratory fitness (VO2peak; male: =55 mL/kg/min; female: 45 mL/kg/min; categorized as =70th percentile by ACSM Guidelines for Exercise Testing and Prescription, 10th Edition; 44, 45, 46, 47)

f.) for female participants, presence of a normal, monthly menstrual cycle with or without prescribed contraceptive methods.

.

Exclusion Criteria:

1. presence of diagnosed cardiovascular, metabolic, or renal disease or dysfunction
2. presence of signs and symptoms suggestive of cardiovascular, metabolic, or renal disease
3. presence of musculoskeletal injury
4. pregnancy
5. history of smoking
6. engagement in an abnormal eating behavior
7. unable to communicate effectively in English
8. moderate cardiorespiratory fitness (VO2peak; male: 46-54 mL/kg/min; female: 36-44 mL/kg/min)
9. elevated or high fasting triglycerides (>150 mg/dL)
10. absence of a normal, monthly menstrual cycle with or without prescribed contraceptive methods

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Fasting triglycerides | Baseline
  Ester derived from glycerol and three fatty acids, representative of the main constituent of body fat in humans.
Post HFM Triglycerides | 4 hours
  Ester derived from glycerol and three fatty acids, representative of the main constituent of body fat in humans.
Fasting total cholesterol | Baseline
  Type of lipid that is required for cell structure, but can contribute to increased risk of heart disease if high due to development of fatty deposits on vascular wall.
Post HFM total cholesterol | 4 hours
  Type of lipid that is required for cell structure, but can contribute to increased risk of heart disease if high due to development of fatty deposits on vascular wall.
Fasting LDL | Baseline
  Low density lipoprotein that transports fat molecules in the body. Associated with high levels of cholesterol.
Post HFM LDL | 4 hours
  Low density lipoprotein that transports fat molecules in the body. Associated with high levels of cholesterol.
Fasting HDL | Baseline
  High density lipoprotein that transports fat molecules in the body. Associated with carrying cholesterol to the liver for degradation.
Post HFM HDL | 4 hours
  High density lipoprotein that transports fat molecules in the body. Associated with carrying cholesterol to the liver for degradation.
Fasting non-HDL | Baseline
  Total cholesterol minus HDL, often associated with a better assessment of risk for heart disease.
Post HFM non-HDL | 4 hours
  Total cholesterol minus HDL, often associated with a better assessment of risk for heart disease.
Fasting LDL/HDL ratio | Baseline
  Assessment of risk for heart disease.
Post HFM LDL/HDL ratio | 4 hours
  Assessment of risk for heart disease.
Fasting anti-inflammatory surface receptor expression | Baseline
  CD14, CD206 - monocyte receptors associated with defining subsets and inflammatory differentiation of macrophages.
Post HFM anti-inflammatory surface receptor expression | 4 hours
  CD14, CD206 - monocyte receptors associated with defining subsets and inflammatory differentiation of macrophages.
Fasting pro-inflammatory surface receptor expression | Baseline
  CD16, CD86 - monocyte receptors associated with defining subsets and inflammatory differentiation of macrophages.
Post HFM pro-inflammatory surface receptor expression | 4 hours
  CD16, CD86 - monocyte receptors associated with defining subsets and inflammatory differentiation of macrophages.
Fasting brachial artery flow-mediated dilation | Baseline
  Dilation of brachial artery when blood flow increases in artery. Measured by non-invasive ultrasound.
Post HFM brachial artery flow-mediated dilation | 5.5 hours
  Dilation of brachial artery when blood flow increases in artery. Measured by non-invasive ultrasound.
Fasting superficial artery flow-mediated dilation | Baseline
  Dilation of superficial artery when blood flow increases in artery. Measured by non-invasive ultrasound.
Post HFM superficial artery flow-mediated dilation | 5.5 hours
  Dilation of superficial artery when blood flow increases in artery. Measured by non-invasive ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Franco, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No